CLINICAL TRIAL: NCT06892314
Title: Association Between CGM Metrics in Type 2 Diabetes Pregnancy and Perinatal Morbidity
Acronym: PREG CGM
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Sud Francilien (Other)
Responsible Party: Sponsor
Other Study IDs: 2025/0006
Record Dates: First submitted 2025-03-13; First posted 2025-03-24 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes Mellitus (T2DM); Pregnancy
Keywords: Type 2 diabetes mellitus; Continuous glucose monitoring; Pregnancy; Retrospective cohort study
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients
  Interventions: Biological: Exposure to hyperglycemia (type 2 diabetes)

INTERVENTIONS:
Biological: Exposure to hyperglycemia (type 2 diabetes) — Exposure to hyperglycemia, in the context of type 2 diabetes, as measured by continuous glucose monitoring

SUMMARY:
The purpose of this observational study is to measure the association between continuous glucose monitoring (CGM) parameters and perinatal morbidity in offspring of women with type 2 diabetes. Specifically, the study will assess whether gestational age interacts with metabolic control in influencing perinatal morbidity, as well as the impact of the timing of CGM initiation during pregnancy.

DETAILED DESCRIPTION:
Continuous glucose monitoring (CGM) data in pregnant women living with type 2 diabetes (T2D) and its association with perinatal morbidity are very recent and remain scarce. Moreover, perinatal morbidity appears to differ in these patients compared to pregnancies affected by type 1 diabetes or gestational diabetes.

As a result, a deeper understanding is needed to identify the most relevant glycemic parameters and, in particular, the gestational age most critical for metabolic control.

Furthermore, uncertainty remains regarding the benefits of early CGM use in this population, which is characterized by early-onset T2D. A description of this population in the French context is therefore of particular interest.

This single-centre observational study will consist of a retrospective cohort of patients with type 2 diabetes and pregnancy with pregnancy follow-up and delivery at the Centre Hospitalier Sud-Francilien between 1 January 2020 and 31 January 2025.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Patient diagnosed with type 2 diabetes before or during pregnancy (fasting blood glucose > 126 mg/dL, blood glucose > 200 mg/dL after an oral glucose tolerance test, or HbA1c > 6.5%)
* Patient who has undergone continuous glucose monitoring at least once during pregnancy

Exclusion Criteria:

* Multiple pregnancy
* Pregnancy terminated before 20 weeks of amenorrhea
* Delivery outside CHSF
* Patient and/or legal guardians of the newborn who objected to the use of data

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient diagnosed with type 2 diabetes before or during pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2025-05-15 (Actual); Primary Completion 2025-11-26 (Actual); Study Completion 2025-11-26 (Actual)

PRIMARY OUTCOMES:
time in range (63-140 mg/dL) in pourcentage | up to delivery
  Correlation between time in range (63-140 mg/dL) during pregnancy and perinatal risk, assessed using a composite outcome including preterm birth, birth weight > 90th percentile for gestational age, neonatal hypoglycemia, shoulder dystocia, neonatal resuscitation, neonatal hyperbilirubinemia, and perinatal mortality.
preterm birth : yes or no | at delivery
  Correlation between time in range (63-140 mg/dL) during pregnancy and perinatal risk, assessed using a composite outcome including preterm birth, birth weight > 90th percentile for gestational age, neonatal hypoglycemia, shoulder dystocia, neonatal resuscitation, neonatal hyperbilirubinemia, and perinatal mortality.
birth weight in kilogramme | at delivery
  Correlation between time in range (63-140 mg/dL) during pregnancy and perinatal risk, assessed using a composite outcome including preterm birth, birth weight > 90th percentile for gestational age, neonatal hypoglycemia, shoulder dystocia, neonatal resuscitation, neonatal hyperbilirubinemia, and perinatal mortality.
neonatal hypoglycemia : yes or no | at delivery
  Correlation between time in range (63-140 mg/dL) during pregnancy and perinatal risk, assessed using a composite outcome including preterm birth, birth weight > 90th percentile for gestational age, neonatal hypoglycemia, shoulder dystocia, neonatal resuscitation, neonatal hyperbilirubinemia, and perinatal mortality.
shoulder dystocia : yes or no | at delivery
  Correlation between time in range (63-140 mg/dL) during pregnancy and perinatal risk, assessed using a composite outcome including preterm birth, birth weight > 90th percentile for gestational age, neonatal hypoglycemia, shoulder dystocia, neonatal resuscitation, neonatal hyperbilirubinemia, and perinatal mortality.
neonatal resuscitation : yes or no | at delivery
  Correlation between time in range (63-140 mg/dL) during pregnancy and perinatal risk, assessed using a composite outcome including preterm birth, birth weight > 90th percentile for gestational age, neonatal hypoglycemia, shoulder dystocia, neonatal resuscitation, neonatal hyperbilirubinemia, and perinatal mortality.
perinatal mortality : yes or no | at delivery
  Correlation between time in range (63-140 mg/dL) during pregnancy and perinatal risk, assessed using a composite outcome including preterm birth, birth weight > 90th percentile for gestational age, neonatal hypoglycemia, shoulder dystocia, neonatal resuscitation, neonatal hyperbilirubinemia, and perinatal mortality.

SECONDARY OUTCOMES:
mean glucose (mmol/L) | up to delivery
  Correlation between characteristics of pregnant patients with T2D and their newborns, including diabetes management and delivery details
time in range (less than 63 mg/dL) in pourcentage | up to delivery
  Correlation between characteristics of pregnant patients with T2D and their newborns, including diabetes management and delivery details
glucose management indicator in pourcentage | up to delivery
  Correlation between distribution of characteristics of pregnant patients with T2D and their newborns, including diabetes management and delivery details
glycemic coefficient of variation in pourcentage | up to delivery
  Correlation between distribution of characteristics of pregnant patients with T2D and their newborns, including diabetes management and delivery details

CONTACTS AND LOCATIONS:
Overall Officials: Coralie AMADOU, MD, Principal Investigator — Centre Hospitalier Sud Francilien
Locations (1):
- Centre Hospitalier Sud Francilien, Corbeil-Essonnes, France, France

IPD SHARING:
Plan to Share IPD: No